CLINICAL TRIAL: NCT03976440
Title: Simplified Regional Citrate Anticoagulation Protocols for CVVH, CVVHDF and SLED Focused on the Prevention of RRT-related Hypophosphatemia and Optimization of Acid-base Balance: a Pilot Study
Brief Title: Simplified Regional Citrate Anticoagulation Protocols for CVVH, CVVHDF and SLED: a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Enrico Fiaccadori, University Professor, University of Parma
Other Study IDs: CRRT/SLED-RCA protocol
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Acute Renal Failure; Dialysis Related Complication; Hypophosphatemia; Hypomagnesemia
Keywords: Acute kidney injury; Regional citrate anticoagulation; Continuous renal replacement therapy; Prolonged intermittent renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Hypophosphatemia | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples to determine the citrate concentration in course of renal replacement therapy (RRT) in the setting of regional citrate anticoagulation (RCA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Renal Replacement Therapy (RRT) start — At the discretion of the nephrologist, treatment modality will be selected among CVVH, CVVHDF or SLED. Whatever the RRT modality, the investigators will adopt RCA as the standard anticoagulation strategy

SUMMARY:
The aim of the study are: 1) To evaluate the occurrence of acid-base alterations and the incidence of hypophosphatemia during different modalities of Renal Replacement Terapy (RRT) in critically ill patients [CVVH, CVVHDF and SLED (Sustained Low-Efficiency Dialysis)] by using a simplified Regional Citrate Anticoagulation (RCA) protocol combined with the adoption of a phosphate-containing solution as dialysate and/or replacement fluid; 2) To optimize the infusion rates of different solutions adopted, including citrate, in order to obtain an appropriate electrolyte and buffer supply. The final aim of this approach will be to reduce the need for frequent monitoring of acid-base status and electrolytes (with special regard to ionized calcium levels), and to avoid the need for frequent adjustments of RCA-RRT parameters (infusion rate of different solutions, electrolytes supplementation in the course of RRT). This approach could allow to simplify anticoagulation protocols with citrate, in order to minimize potential concerns hampering a wider diffusion of RCA in daily practice.

DETAILED DESCRIPTION:
The need for continuous anticoagulation represents a potential drawback of RRT modalities. KDIGO 2012 guidelines on acute kidney injury (AKI) suggest the adoption of RCA as first choice anticoagulation modality for continuous RRT (CRRT) in patients without contraindications for citrate. Citrate has been also introduced as anticoagulant for SLED and its use in the context of a mainly diffusive prolonged intermittent modality has been shown to represent an easy and safe method to maintain the extracorporeal circuit when concentrated citrate solutions, such as ACD-A are used. Hypophosphatemia is a known issue of RRT, and has been reported in up to 50-80% of cases when standard RRT solutions are used, especially in continuous/prolonged intermitted modalities when high RRT doses are delivered. RRT-related phosphate depletion should be avoided in critically ill patients due to the relevant hypophosphatemia-associated complications in this clinical setting. The adoption of phosphate-containing CRRT solutions could reduce the incidence of hypophosphatemia and minimize the need for parenteral phosphorus supplementation.The adoption of a commercially available phosphate-containing CRRT solution, in the setting of RCA-RRT may allow to meet the double target of minimizing RRT-induced hypophosphatemia and ensuring an adequate circuit life, also avoiding electrolyte and acid-base derangements.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* critically ill patients requiring continuous or prolonged intermittent renal replacement therapy for severe acute kidney injury (AKI)
* critically ill patients requiring continuous or prolonged intermittent renal replacement therapy for end stage renal disease (ESRD)

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients aged >=18 years with severe acute kidney injury (AKI) or end stage renal disease (ESRD) requiring renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Hypophosphatemia | 72 hours
  Occurrence of hypophosphatemia during the first 72 hours of continuous renal replacement therapy (CRRT) or sustained low-efficiency dialysis (SLED)
Acid-base derangements | 72 hours
  Occurrence of acid-base derangements during CRRT and SLED using a simplified RCA protocol
Variations of RCA-RRT parameters | 72 hours
  Evaluation of the need for variations of RCA-RRT dialysis parameters from initial RRT settings
Variations of RCA-RRT solutions | 72 hours
  Evaluation of the need for variations in RRT solutions flow rate rom initial RRT settings

SECONDARY OUTCOMES:
Hypomagnesemia | 72 hours
  Occurrence of hypomagnesemia during the first 72 hours of CRRT or SLED
Efficacy of RCA | 72 hours
  Efficacy of RCA in terms of circuit lifetime and filter efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma - UO Nefrologia AOU, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fliser D, Kielstein JT. Technology Insight: treatment of renal failure in the intensive care unit with extended dialysis. Nat Clin Pract Nephrol. 2006 Jan;2(1):32-9. doi: 10.1038/ncpneph0060. PMID 16932387
- [Result] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Result] Mariano F, Pozzato M, Canepari G, Vitale C, Bermond F, Sacco C, Amore A, Manes M, Navino C; Piedmont and Aosta Valley Section of Italian Society of Nephrology. Renal replacement therapy in intensive care units: a survey of nephrological practice in northwest Italy. J Nephrol. 2011 Mar-Apr;24(2):165-76. doi: 10.5301/jn.2010.2380. PMID 20586025
- [Result] Marshall MR, Golper TA. Low-efficiency acute renal replacement therapy: role in acute kidney injury. Semin Dial. 2011 Mar-Apr;24(2):142-8. doi: 10.1111/j.1525-139X.2011.00829.x. PMID 21517979
- [Result] Marshall MR, Creamer JM, Foster M, Ma TM, Mann SL, Fiaccadori E, Maggiore U, Richards B, Wilson VL, Williams AB, Rankin AP. Mortality rate comparison after switching from continuous to prolonged intermittent renal replacement for acute kidney injury in three intensive care units from different countries. Nephrol Dial Transplant. 2011 Jul;26(7):2169-75. doi: 10.1093/ndt/gfq694. Epub 2010 Nov 12. PMID 21075821
- [Result] Schwenger V, Weigand MA, Hoffmann O, Dikow R, Kihm LP, Seckinger J, Miftari N, Schaier M, Hofer S, Haar C, Nawroth PP, Zeier M, Martin E, Morath C. Sustained low efficiency dialysis using a single-pass batch system in acute kidney injury - a randomized interventional trial: the REnal Replacement Therapy Study in Intensive Care Unit PatiEnts. Crit Care. 2012 Jul 27;16(4):R140. doi: 10.1186/cc11445. PMID 22839577
- [Result] Fieghen HE, Friedrich JO, Burns KE, Nisenbaum R, Adhikari NK, Hladunewich MA, Lapinsky SE, Richardson RM, Wald R; University of Toronto Acute Kidney Injury Research Group. The hemodynamic tolerability and feasibility of sustained low efficiency dialysis in the management of critically ill patients with acute kidney injury. BMC Nephrol. 2010 Nov 25;11:32. doi: 10.1186/1471-2369-11-32. PMID 21106112
- [Result] Kron J, Kron S, Wenkel R, Schuhmacher HU, Thieme U, Leimbach T, Kern H, Neumayer HH, Slowinski T. Extended daily on-line high-volume haemodiafiltration in septic multiple organ failure: a well-tolerated and feasible procedure. Nephrol Dial Transplant. 2012 Jan;27(1):146-52. doi: 10.1093/ndt/gfr269. Epub 2011 May 28. PMID 21622989
- [Result] Kielstein JT, Kretschmer U, Ernst T, Hafer C, Bahr MJ, Haller H, Fliser D. Efficacy and cardiovascular tolerability of extended dialysis in critically ill patients: a randomized controlled study. Am J Kidney Dis. 2004 Feb;43(2):342-9. doi: 10.1053/j.ajkd.2003.10.021. PMID 14750100
- [Result] Fiaccadori E, Maggiore U, Parenti E, Giacosa R, Picetti E, Rotelli C, Tagliavini D, Cabassi A. Sustained low-efficiency dialysis (SLED) with prostacyclin in critically ill patients with acute renal failure. Nephrol Dial Transplant. 2007 Feb;22(2):529-37. doi: 10.1093/ndt/gfl627. Epub 2006 Oct 28. PMID 17071958
- [Result] Fiaccadori E, Regolisti G, Cademartiri C, Cabassi A, Picetti E, Barbagallo M, Gherli T, Castellano G, Morabito S, Maggiore U. Efficacy and safety of a citrate-based protocol for sustained low-efficiency dialysis in AKI using standard dialysis equipment. Clin J Am Soc Nephrol. 2013 Oct;8(10):1670-8. doi: 10.2215/CJN.00510113. Epub 2013 Aug 29. PMID 23990164
- [Result] Morabito S, Pistolesi V, Tritapepe L, Fiaccadori E. Regional citrate anticoagulation for RRTs in critically ill patients with AKI. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2173-88. doi: 10.2215/CJN.01280214. Epub 2014 Jul 3. PMID 24993448
- [Result] Fiaccadori E, Maggiore U, Clima B, Melfa L, Rotelli C, Borghetti A. Incidence, risk factors, and prognosis of gastrointestinal hemorrhage complicating acute renal failure. Kidney Int. 2001 Apr;59(4):1510-9. doi: 10.1046/j.1523-1755.2001.0590041510.x. PMID 11260415
- [Result] Fiaccadori E, Pistolesi V, Mariano F, Mancini E, Canepari G, Inguaggiato P, Pozzato M, Morabito S. Regional citrate anticoagulation for renal replacement therapies in patients with acute kidney injury: a position statement of the Work Group "Renal Replacement Therapies in Critically Ill Patients" of the Italian Society of Nephrology. J Nephrol. 2015 Apr;28(2):151-64. doi: 10.1007/s40620-014-0160-2. Epub 2015 Jan 14. PMID 25585821
- [Result] Bellomo R, Kellum JA, Ronco C. Acute kidney injury. Lancet. 2012 Aug 25;380(9843):756-66. doi: 10.1016/S0140-6736(11)61454-2. Epub 2012 May 21. PMID 22617274
- [Result] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Result] Hsu CY, McCulloch CE, Fan D, Ordonez JD, Chertow GM, Go AS. Community-based incidence of acute renal failure. Kidney Int. 2007 Jul;72(2):208-12. doi: 10.1038/sj.ki.5002297. Epub 2007 May 16. PMID 17507907
- [Result] Bagshaw SM, George C, Bellomo R; ANZICS Database Management Committee. Early acute kidney injury and sepsis: a multicentre evaluation. Crit Care. 2008;12(2):R47. doi: 10.1186/cc6863. Epub 2008 Apr 10. PMID 18402655
- [Result] Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA. RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. Crit Care. 2006;10(3):R73. doi: 10.1186/cc4915. Epub 2006 May 12. PMID 16696865
- [Result] Morabito S, Pistolesi V, Cibelli L, Pierucci A. [Continuous renal replacement therapies (CRRT) will remain the most widely adopted dialysis modality in the critically ill]. G Ital Nefrol. 2009 Jan-Feb;26(1):13-21. Italian. PMID 19255959
- [Result] Brophy PD, Somers MJ, Baum MA, Symons JM, McAfee N, Fortenberry JD, Rogers K, Barnett J, Blowey D, Baker C, Bunchman TE, Goldstein SL. Multi-centre evaluation of anticoagulation in patients receiving continuous renal replacement therapy (CRRT). Nephrol Dial Transplant. 2005 Jul;20(7):1416-21. doi: 10.1093/ndt/gfh817. Epub 2005 Apr 26. PMID 15855212
- [Result] Oudemans-van Straaten HM, Wester JPJ, de Pont ACJM, Schetz MRC. Anticoagulation strategies in continuous renal replacement therapy: can the choice be evidence based? Intensive Care Med. 2006 Feb;32(2):188-202. doi: 10.1007/s00134-005-0044-y. Epub 2006 Feb 2. PMID 16453140
- [Result] Tolwani AJ, Wille KM. Anticoagulation for continuous renal replacement therapy. Semin Dial. 2009 Mar-Apr;22(2):141-5. doi: 10.1111/j.1525-139X.2008.00545.x. PMID 19426417
- [Result] Mariano F. [Citrate: a different mental approach to extracorporeal circuit anticoagulation]. G Ital Nefrol. 2012 Jan-Feb;29(1):27-32. Italian. PMID 22388903
- [Result] Mariano F, Triolo G. [Anticoagulation of extracorporeal circuit in critically ill patients]. G Ital Nefrol. 2007 Jan-Feb;24(1):34-42. Italian. PMID 17342691
- [Result] Oudemans-van Straaten HM. Citrate anticoagulation for continuous renal replacement therapy in the critically ill. Blood Purif. 2010;29(2):191-6. doi: 10.1159/000245646. Epub 2010 Jan 8. PMID 20093826
- [Result] Davenport A, Tolwani A. Citrate anticoagulation for continuous renal replacement therapy (CRRT) in patients with acute kidney injury admitted to the intensive care unit. NDT Plus. 2009 Dec;2(6):439-47. doi: 10.1093/ndtplus/sfp136. Epub 2009 Sep 25. PMID 25949376
- [Result] Mariano F, Tedeschi L, Morselli M, Stella M, Triolo G. Normal citratemia and metabolic tolerance of citrate anticoagulation for hemodiafiltration in severe septic shock burn patients. Intensive Care Med. 2010 Oct;36(10):1735-1743. doi: 10.1007/s00134-010-1909-2. Epub 2010 May 18. PMID 20480135
- [Result] Chadha V, Garg U, Warady BA, Alon US. Citrate clearance in children receiving continuous venovenous renal replacement therapy. Pediatr Nephrol. 2002 Oct;17(10):819-24. doi: 10.1007/s00467-002-0963-6. Epub 2002 Sep 7. PMID 12376810
- [Result] Mariano F, Tetta C, Stella M, Biolino P, Miletto A, Triolo G. Regional citrate anticoagulation in critically ill patients treated with plasma filtration and adsorption. Blood Purif. 2004;22(3):313-9. doi: 10.1159/000078788. PMID 15256798
- [Result] Hetzel GR, Taskaya G, Sucker C, Hennersdorf M, Grabensee B, Schmitz M. Citrate plasma levels in patients under regional anticoagulation in continuous venovenous hemofiltration. Am J Kidney Dis. 2006 Nov;48(5):806-11. doi: 10.1053/j.ajkd.2006.07.016. PMID 17060000
- [Result] Mariano F, Morselli M, Bergamo D, Hollo Z, Scella S, Maio M, Tetta C, Dellavalle A, Stella M, Triolo G. Blood and ultrafiltrate dosage of citrate as a useful and routine tool during continuous venovenous haemodiafiltration in septic shock patients. Nephrol Dial Transplant. 2011 Dec;26(12):3882-8. doi: 10.1093/ndt/gfr106. Epub 2011 Mar 8. PMID 21385861
- [Result] Bakker AJ, Boerma EC, Keidel H, Kingma P, van der Voort PH. Detection of citrate overdose in critically ill patients on citrate-anticoagulated venovenous haemofiltration: use of ionised and total/ionised calcium. Clin Chem Lab Med. 2006;44(8):962-6. doi: 10.1515/CCLM.2006.164. PMID 16879061
- [Result] Fukuda T, Toyoshima S, Nakashima Y, Koshitani O, Kawaguchi Y, Momii A. Tolerable infusion rate of citrate based on clinical signs and the electrocardiogram in conscious dogs. Clin Nutr. 2006 Dec;25(6):984-93. doi: 10.1016/j.clnu.2006.01.011. Epub 2006 May 15. PMID 16698131
- [Result] Forsythe RM, Wessel CB, Billiar TR, Angus DC, Rosengart MR. Parenteral calcium for intensive care unit patients. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006163. doi: 10.1002/14651858.CD006163.pub2. PMID 18843706
- [Result] Pozzato M. [Citrate: an additional resource for anticoagulation in continuous replacement therapy]. G Ital Nefrol. 2012 Jan-Feb;29(1):20-6. Italian. PMID 22388902
- [Result] Bai M, Zhou M, He L, Ma F, Li Y, Yu Y, Wang P, Li L, Jing R, Zhao L, Sun S. Citrate versus heparin anticoagulation for continuous renal replacement therapy: an updated meta-analysis of RCTs. Intensive Care Med. 2015 Dec;41(12):2098-110. doi: 10.1007/s00134-015-4099-0. PMID 26482411
- [Result] Monchi M, Berghmans D, Ledoux D, Canivet JL, Dubois B, Damas P. Citrate vs. heparin for anticoagulation in continuous venovenous hemofiltration: a prospective randomized study. Intensive Care Med. 2004 Feb;30(2):260-265. doi: 10.1007/s00134-003-2047-x. Epub 2003 Nov 5. PMID 14600809
- [Result] Hetzel GR, Schmitz M, Wissing H, Ries W, Schott G, Heering PJ, Isgro F, Kribben A, Himmele R, Grabensee B, Rump LC. Regional citrate versus systemic heparin for anticoagulation in critically ill patients on continuous venovenous haemofiltration: a prospective randomized multicentre trial. Nephrol Dial Transplant. 2011 Jan;26(1):232-9. doi: 10.1093/ndt/gfq575. Epub 2010 Sep 27. PMID 20876598
- [Result] Mariano F, Bergamo D, Gangemi EN, Hollo' Z, Stella M, Triolo G. Citrate anticoagulation for continuous renal replacement therapy in critically ill patients: success and limits. Int J Nephrol. 2011;2011:748320. doi: 10.4061/2011/748320. Epub 2011 Mar 16. PMID 21603110
- [Result] Liangos O, Wald R, O'Bell JW, Price L, Pereira BJ, Jaber BL. Epidemiology and outcomes of acute renal failure in hospitalized patients: a national survey. Clin J Am Soc Nephrol. 2006 Jan;1(1):43-51. doi: 10.2215/CJN.00220605. Epub 2005 Oct 26. PMID 17699189
- [Result] Gabutti L, Marone C, Colucci G, Duchini F, Schonholzer C. Citrate anticoagulation in continuous venovenous hemodiafiltration: a metabolic challenge. Intensive Care Med. 2002 Oct;28(10):1419-25. doi: 10.1007/s00134-002-1443-y. Epub 2002 Sep 6. PMID 12373466
- [Result] Oudemans-van Straaten HM, Bosman RJ, Koopmans M, van der Voort PH, Wester JP, van der Spoel JI, Dijksman LM, Zandstra DF. Citrate anticoagulation for continuous venovenous hemofiltration. Crit Care Med. 2009 Feb;37(2):545-52. doi: 10.1097/CCM.0b013e3181953c5e. PMID 19114912
- [Result] Oudemans-van Straaten HM, Kellum JA, Bellomo R. Clinical review: anticoagulation for continuous renal replacement therapy--heparin or citrate? Crit Care. 2011 Jan 24;15(1):202. doi: 10.1186/cc9358. PMID 21345279
- [Result] Palsson R, Niles JL. Regional citrate anticoagulation in continuous venovenous hemofiltration in critically ill patients with a high risk of bleeding. Kidney Int. 1999 May;55(5):1991-7. doi: 10.1046/j.1523-1755.1999.00444.x. PMID 10231464
- [Result] Cassina T, Mauri R, Engeler A, Giannini O. Continuous veno-venous hemofiltration with regional citrate anticoagulation: a four-year single-center experience. Int J Artif Organs. 2008 Nov;31(11):937-43. doi: 10.1177/039139880803101103. PMID 19089795
- [Result] Tolwani AJ, Campbell RC, Schenk MB, Allon M, Warnock DG. Simplified citrate anticoagulation for continuous renal replacement therapy. Kidney Int. 2001 Jul;60(1):370-4. doi: 10.1046/j.1523-1755.2001.00809.x. PMID 11422774
- [Result] Dorval M, Madore F, Courteau S, Leblanc M. A novel citrate anticoagulation regimen for continuous venovenous hemodiafiltration. Intensive Care Med. 2003 Jul;29(7):1186-9. doi: 10.1007/s00134-003-1801-4. Epub 2003 May 22. PMID 12761615
- [Result] Mitchell A, Daul AE, Beiderlinden M, Schafers RF, Heemann U, Kribben A, Peters J, Philipp T, Wenzel RR. A new system for regional citrate anticoagulation in continuous venovenous hemodialysis (CVVHD). Clin Nephrol. 2003 Feb;59(2):106-14. doi: 10.5414/cnp59106. PMID 12608553
- [Result] Buturovic-Ponikvar J, Gubensek J, Ponikvar R. Citrate anticoagulation for postdilutional online hemodiafiltration with calcium-containing dialysate and infusate: significant clotting in the venous bubble trap. Int J Artif Organs. 2008 Apr;31(4):323-8. doi: 10.1177/039139880803100408. PMID 18432588
- [Result] Yang Y, Zhang P, Cui Y, Lang X, Yuan J, Jiang H, Lei W, Lv R, Zhu Y, Lai E, Chen J. Hypophosphatemia during continuous veno-venous hemofiltration is associated with mortality in critically ill patients with acute kidney injury. Crit Care. 2013 Sep 19;17(5):R205. doi: 10.1186/cc12900. PMID 24050634
- [Result] Demirjian S, Teo BW, Guzman JA, Heyka RJ, Paganini EP, Fissell WH, Schold JD, Schreiber MJ. Hypophosphatemia during continuous hemodialysis is associated with prolonged respiratory failure in patients with acute kidney injury. Nephrol Dial Transplant. 2011 Nov;26(11):3508-14. doi: 10.1093/ndt/gfr075. Epub 2011 Mar 7. PMID 21382993
- [Result] Pistolesi V, Zeppilli L, Polistena F, Sacco MI, Pierucci A, Tritapepe L, Regolisti G, Fiaccadori E, Morabito S. Preventing Continuous Renal Replacement Therapy-Induced Hypophosphatemia: An Extended Clinical Experience with a Phosphate-Containing Solution in the Setting of Regional Citrate Anticoagulation. Blood Purif. 2017;44(1):8-15. doi: 10.1159/000453443. Epub 2017 Feb 21. PMID 28219057
- [Derived] Di Mario F, Sabatino A, Regolisti G, Pacchiarini MC, Greco P, Maccari C, Vizzini G, Italiano C, Pistolesi V, Morabito S, Fiaccadori E. Simplified regional citrate anticoagulation protocol for CVVH, CVVHDF and SLED focused on the prevention of KRT-related hypophosphatemia while optimizing acid-base balance. Nephrol Dial Transplant. 2023 Sep 29;38(10):2298-2309. doi: 10.1093/ndt/gfad068. PMID 37037771
- See also: KDIGO Clinical Practice Guideline for Acute Kidney Injury — https://kdigo.org/wp-content/uploads/2016/10/KDIGO-2012-AKI-Guideline-English.pdf